CLINICAL TRIAL: NCT00232817
Title: Intranasal Nicotine for Postoperative Pain Treatment: A Comparison of Its Effects in the Context of Isoflurane-induced Anesthesia Versus Propofol Anesthesia
Brief Title: Anesthesia and Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAA6698
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nicotine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Propofol anesthetic with and without nicotine
  Interventions: Drug: Nicotine (drug)
- 2 (Experimental): isoflurane anesthetic with and without nicotine
  Interventions: Drug: Nicotine (drug)

INTERVENTIONS:
Drug: Nicotine (drug) — nicotine nasal spray (3mg) before surgery

SUMMARY:
The purpose of this study is to compare post-operative pain after anesthesia with either isoflurane or propofol. Each group will be further randomized to receive intranasal nicotine or placebo in order to detect potential pronociceptive action of isoflurane.

The study is a randomized, prospective, double-blinded controlled trial. Eighty adult women undergoing uterine surgery will be recruited for this study. Enrollment in this study is limited to women, because the animal studies suggest that females have a greater hyperalgesic response to volatile anesthetics than do males.

The patient will be given one of two standard anesthetics for their surgery: isoflurane or propofol. The investigators are interested in these two anesthetics because we seek to see if there exists a difference in their effects on a patient's perception of pain, as has been shown to be the case in animal studies but has not yet been studied in humans.

DETAILED DESCRIPTION:
A. Study Proposal and Rational

The purpose of this study is to determine whether intranasal nicotine can decrease the negative side effects of the general anesthetic isoflurane. Isoflurane and other volatile anesthetics are potent antagonists of central nicotinic receptors. Nicotinic receptors are inhibited by isoflurane at the low concentrations that are present on emergence from anesthesia. Evidence from animal experiments suggests that inhibition of nicotinic receptors may cause increased sensitivity to pain and amnesia that occurs at low anesthetic concentrations. These anesthetic concentrations are frequently present on emergence from anesthesia. In these experiments, treatment with nicotine prevented the hyperalgesic state caused by isoflurane.

Intranasal nicotine treatment has been used in smokers as an aid to smoking cessation. As nicotine acts as an agonist at sympathetic ganglia, it can cause increases in heart rate and blood pressure. At the dose to be used in this protocol (3mg intranasally) there was an average increase of 7 mM of mercury in systolic blood pressure and no change in diastolic blood pressure or heart rate in nonsmoking volunteers.

B. Study Design and Statistical Analysis

The study is a randomized prospective controlled trial. Women scheduled to undergo total abdominal hysterectomy or myomectomy will be randomly allocated intranasal nicotine or intranasal saline before emergence from a standard general anesthetic. The patient will be randomized to one of two standard anesthetics regimens that are described below. Both patient and investigator will be blinded to treatment. Nicotine or saline will be placed in a single use nasal spray bottle by the research pharmacy and identified by number. Randomization will be accomplished with a random number table. Patients will be enrolled sequentially.

The study wishes to detect a 50% change in pain sensitivity and in our other studies, Visual Analog Pain Scale (VAS) scores and patient-controlled analgesia (PCA) utilization varied by approximately 40% (pooled variance). In order to achieve 80% power and p<0.05, 40 women per group will be enrolled (total of 80 women). This study will include only female patients as animal studies suggest that females have a greater hyperalgesic response to isoflurane than males. Patients treated with nicotine will be compared to those treated with placebo for VAS score, PCA utilization and memory at 1 and 24 hours.

C. Study Procedure

The study subjects will be given one of two standardized anesthetics by an anesthesiologist at New York Presbyterian Hospital (NYPH) not involved with the study. The anesthesiologist will be familiarized with the study protocol prior to the surgery. The anesthetic protocols chosen are typical for this type of surgery, but is standardized to decrease variability in postoperative condition.

After placing an intravenous catheter and standard anesthetic monitors, the patient will be pre oxygenated. Fentanyl will be administered at 12 micrograms/kg and a continuous infusion of 12 micrograms/kg/hr will be begun. Vecuronium 1 mg will be used to reduce fasciculation from succinylcholine. Anesthesia will be induced with propofol 2 mg/kg and intubation facilitated with succinylcholine 12 mg/kg. Anesthesia will be maintained with either isoflurane or propofol titrated by the anesthesiologist. All patients will be have a BIS monitor (a measure of processed EEG) titrated between 45-60 to assure adequacy and equivalence of anesthesia. Hypotension will be treated with ephedrine or phenylephrine as deemed necessary by the anesthesiologist. Hypertension will be treated with hydralazine or labatelol in doses determined by the anesthesiologist. If other hemodynamic or anesthetic drugs are deemed necessary by the anesthesiologist, the patient will be removed from the protocol.

After closure of the abdominal fascia (typically, approximately 5 minutes before anticipated completion of the surgery) the general anesthetic and fentanyl drip will be titrated to off. Muscle relaxant will be reversed with neostigmine 0.1 mg/kg and glycopyrolate 0.01 mg/kg. At this time the study drug (nicotine 3 mg or saline) will be administered intranasally 3 mg (half to each nostril). The patient will be extubated by the anesthesiologist when she meets normal criteria (as determined by the anesthesiologist).

Five minutes after extubation, the patient will be asked for a VAS score by the study coordinator. Pain will be treated with fentanyl by the anesthesiologist, 1 mg/kg every 5 minutes until VAS score is less than 3. PCA will then be begun with morphine 1 mg with a lockout of 6 minutes and a maximal 1 hour dose of 10 mg. A rescue dose of 3 mg morphine will be available to be administered by the nurse through the PCA every 5 minutes for a maximum of 12 mg in 4 hours. If pain is inadequately treated there will be an option to increase the patient demand dose to 1.5 mg morphine and the 1 hour maximum to 15 mg. This is a typical PCA protocol for this surgery.

Post-anesthesia care unit (PACU) monitoring will be standard except that the patient's pain intensity will be monitored every 5 minutes in the first hour, once at the second hour and once at the twenty four hour period postoperatively by the study coordinator who will ask for a VAS score. PCA utilization will be determined from the amount of narcotic used from the PCA machine. The study will last during the patient's first postoperative day.

D. Study Drugs

Nicotine has been used commonly on an outpatient basis for smoking cessation. The investigators have chosen the intranasal route because of the kinetics of its action. Intranasal nicotine has its peak effect in five minutes and is dissipated in about 1 hour. In human studies, the hyperalgesic effect after a volatile anesthetic lasted about 1 hour.

As nicotine acts as an agonist at sympathetic ganglia, it can cause increases in heart rate and blood pressure. At the dose to be used in this protocol (3mg intranasally) there was an average increase of 7 mM of mercury in systolic blood pressure and no change in diastolic blood pressure or heart rate in nonsmoking volunteers. The preliminary data do not show any significant increase in blood pressure or heart rate in patients who received nicotine.

The investigators have chosen to study a dose of 3 mg because that dose had minimal hemodynamic effects and resulted in an arterial peak concentration of 100 microM and a steady state venous concentration of 30 microM nicotine. As nicotine crosses the blood brain barrier, these concentrations would be expected to result in significant activation of nicotinic receptors in the brain and spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* female sex
* present to New York Presbyterian Hospital for open pelvic surgery

Exclusion Criteria:

* smoking
* uncontrolled hypertension
* myocardial disease
* history of stroke

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2005-07 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela D Flood, M.D., Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Background] Fishbein L, O'Brien P, Hutson A, Theriaque D, Stacpoole PW, Flotte T. Pharmacokinetics and pharmacodynamic effects of nicotine nasal spray devices on cardiovascular and pulmonary function. J Investig Med. 2000 Nov;48(6):435-40. PMID 11094866
- [Background] Flood P, Ramirez-Latorre J, Role L. Alpha 4 beta 2 neuronal nicotinic acetylcholine receptors in the central nervous system are inhibited by isoflurane and propofol, but alpha 7-type nicotinic acetylcholine receptors are unaffected. Anesthesiology. 1997 Apr;86(4):859-65. doi: 10.1097/00000542-199704000-00016. PMID 9105230
- [Background] Flood P, Sonner JM, Gong D, Coates KM. Isoflurane hyperalgesia is modulated by nicotinic inhibition. Anesthesiology. 2002 Jul;97(1):192-8. doi: 10.1097/00000542-200207000-00027. PMID 12131122
- [Background] Guthrie SK, Zubieta JK, Ohl L, Ni L, Koeppe RA, Minoshima S, Domino EF. Arterial/venous plasma nicotine concentrations following nicotine nasal spray. Eur J Clin Pharmacol. 1999 Nov;55(9):639-43. doi: 10.1007/s002280050686. PMID 10638392
- [Background] Violet JM, Downie DL, Nakisa RC, Lieb WR, Franks NP. Differential sensitivities of mammalian neuronal and muscle nicotinic acetylcholine receptors to general anesthetics. Anesthesiology. 1997 Apr;86(4):866-74. doi: 10.1097/00000542-199704000-00017. PMID 9105231
- [Background] Zhang Y, Eger EI 2nd, Dutton RC, Sonner JM. Inhaled anesthetics have hyperalgesic effects at 0.1 minimum alveolar anesthetic concentration. Anesth Analg. 2000 Aug;91(2):462-6. doi: 10.1097/00000539-200008000-00044. PMID 10910869
- [Background] Flood P, Daniel D. Intranasal nicotine for postoperative pain treatment. Anesthesiology. 2004 Dec;101(6):1417-21. doi: 10.1097/00000542-200412000-00023. PMID 15564950

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine: Patients were administered anesthetic (1-2 μg/kg fentanyl and 1 mg vecuronium) before surgery. After surgery, patients were administered with a nicotine nasal spray (3 mg Nicotrol).
- Placebo: Patients were administered anesthetic (1-2 μg/kg fentanyl and 1 mg vecuronium) before surgery. After surgery, patients were administered with a saline nasal spray.
Period: Overall Study
Arm/Group | Nicotine | Placebo
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment - Nicotine: Nicotine nasal spray
- Treatment - Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Treatment - Nicotine | Treatment - Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (9.2) | 46.1 (6.9) | 44.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Country
  Participants
    United States | 10 | 10 | 20
Weight [Mean (Standard Deviation); unit: pounds] — Pounds Population: no difference
  pounds | 143.5 (37.0) | 146.3 (29.0) | 145.0 (32.4)

OUTCOME MEASURES:

1. Primary Outcome: Score on a Pain Rating Scale (Numerical Analog Score)
Description: Pain was reported on the Numerical Rating Scale for pain (NRS) with 0=no pain and 10=worst pain. Pain was assessed at 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 120, and 1440 minutes post-op, and the average of all time-points is reported.
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 10 | 10
scores on a scale | 1.5 (0.5) | 4.9 (1.4)

2. Secondary Outcome: Cumulative Morphine Usage
Description: The amount of morphine used by each patient at the following time points will be summed: 5, 10, 15, 20, 25, 30, 35, 40, 45, 60, 120, and 1440 minutes post-operative. A patient-controlled analgesia pump was programmed to deliver a dose of 1 mg morphine when the button is pressed with a lockout interval of 6 min and a maximal dose during 1 h of 10 mg. The pump is also programmed to allow a rescue dose of 3mg morphine to be administered by a nurse every 5 min with additional 12 mg morphine maximally by this route every 4 hours. A patient could receive 24 mg of morphine as a maximal dose in the first hour.
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Nicotine; Placebo: Treatment
Arm/Group | Nicotine | Placebo
Number analyzed (Participants) | 10 | 10
mg | 35.3 (23.7) | 51.6 (26.6)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Nicotine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No